CLINICAL TRIAL: NCT01918384
Title: Phase II Study of Nonsense Readthrough Compound NPC-14 (Arbekacin Sulfate) to Explore Safety, Tolerability, and Efficacy in Duchenne Muscular Dystrophy Patients (NORTH POLE DMD Study)
Brief Title: Phase II Study of NPC-14 (Arbekacin Sulfate) to Explore Safety, Tolerability, and Efficacy in Duchenne Muscular Dystrophy
Acronym: NORTH POLE DMD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kobe University (Industry)
Collaborators: Japan Medical Association (Industry); Nobelpharma (Industry)
Responsible Party: Principal Investigator, Yasuhiro Takeshima, MD, PhD, Kobe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPC-14-1; JMA-IIA00134 (Other: Center for clinical trials, Japan Medical Association)
Record Dates: First submitted 2013-08-01; First posted 2013-08-07 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne muscular dystrophy; NPC-14; Arbekacin; nonsense; readthrough
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — arbekacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPC-14 (Experimental): Intravenous drip, QW, 36 weeks, Dose will be adjusted and maintained by therapeutic drug monitoring of peak serum levels of NPC-14
  Interventions: Drug: NPC-14
- Placebo (Placebo Comparator): Dose will be adjusted by volume of distribution (Vd) of patients in accordance with the NPC-14 dose regimen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPC-14 — NPC-14 will be administrated as following steps. The dose of NPC-14 will be calculated and adjusted by a non-blinded medical doctor and/or a non-blinded pharmacist.
  * An initial dose of NPC-14 will be half of that calculated by distribution volume：Vd based on patient age for safety reason.
  * After the initial administration, the dose of NPC-14 will be adjusted and maintained by actual Vd, therapeutic drug monitoring of peak serum levels of NPC-14
  Other Names: Arbekacin
  Arms: NPC-14
Drug: Placebo — Dose will be adjusted by volume of distribution (Vd) of patients in accordance with the NPC-14 dose regimen
  Arms: Placebo

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is inherited neuromuscular disorders due to mutation in the gene that encodes critical muscle protein called dystrophin. Currently, there is no effective treatment option for the disease. A pharmacological approach by promoting mRNA translation regardless of the presence of premature stop codons by nonsense mutation, called the readthrough strategy, has been developing recently for DMD with nonsense mutation. NPC-14 is a candidate compound for the readthrough strategy, since effective readthrough activities were demonstrated in nonclinical studies. This study is a phase II study designed to assess safety, tolerability, and efficacy of NPC-14 in ambulant DMD patients with nonsense mutation that were confirmed by whole genome analysis. These goals will be accomplished by monitoring adverse events by physical examination, cardiac, pulmonary, auditory, balance, and laboratory tests as safety endpoints, and dystrophin expression in muscle biopsy as primary efficacy endpoint, muscle function (NSAA, timed test, muscle strength (QMT, MMT) , dairy activities by lifecorder), and biomarkers as secondary efficacy endpoints. The study is a randomized, double blind, placebo-controlled study in 21 DMD patients. After screening, eligible patients are allocated dynamically to weekly NPC-14 or a placebo (saline) in a 2:1 ratio and will receive study drugs for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DMD resulting from a nonsense mutation by whole genome sequencing of the dystrophin gene
2. To have intact right or left biceps muscles, or an alternative muscle group that is able to be underwent for appropriate evaluation of efficacy
3. To meet the following criteria at screening (baseline visit), within 30 days prior to the first dose of study drug

   * Ambulant and able to walk at least 75 meters during the 6MWT
   * Able to comply with and complete all protocol requirements, and judged by the investigator to be appropriate to participate in the study from the screening results
4. Aged at least 4 years at the time of giving informed consent
5. Male
6. Able to be hospitalized for the study requirement
7. Signed Informed consent by parents/legal guardian and/or signed assent by the subject (age of assent to be determined by IRB)

Exclusion Criteria:

1. Prior exposure to investigational medicines that have a potential of restoring dystrophin or other functional protein (readthrough, exon skipping, utrophin upregulation therapy etc.)
2. Known mutation at nucleotide 1555 in 12S rRNA gene of mitochondrial DNA, and/or personally or families have been treated or have a history of eight cranial nerve disorder （hearing loss、vertigo、tinnitus etc.）as a result of aminoglycoside use
3. Inability to hear within the range of 0 to 25 dB by pure tone audiometry, abnormalities on auditory brainstem response audiometry, and/or loss of frequency by distortion product oto acoustic emissions at screening
4. Poor oral intake or enable to oral intake, and/or bad general status
5. Known allergies to NPC-14, other aminoglycosides, and/or bacitracin
6. Presence of anti-dystrophin antibody at the baseline assessments
7. Cys-C ≥1.2 mg/L and/or creatinine concentration >1.5 times the upper limit of age corrected normal range
8. Left ventricular ejection fraction (EF) <40% or left ventricular fractional shortening (FS) <25%, and/or ≥480 msec QTc (corrected QT interval by Fridericia's method)
9. Need of mechanical ventilation
10. Forced vital capacity (FVC) <50% predicted
11. Clinically significant concomitant diseases (hematology, psychoneurotic, hepatic, pulmonary, endocrine, immune, renal, and gastroenterological diseases), and/or cancer
12. Impairment of intellectual functions, and/or expressive language ability which might interfere with study assessments
13. Treatment with other systemic aminoglycoside within 6 months prior to the first administration of study drug
14. Initiation of systemic glucocorticosteroids treatment, and/or start exercise cure, physical therapy, or occupational therapy which might interfere with study assessments. Changing of dose and schedule of systemic glucocorticosteroids within 6 months prior to the first administration of study drug
15. History of any surgical procedure within months prior to the first administration of study drug or have a plan during study
16. History of sever allergy from food and medicine like an anaphylaxis shock or generalized rash
17. Participation in any other clinical trial and intake of any investigational drug within 6month of study entry

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability (Adverse events) | Up to 38 weeks (36 weeks treatment period and 2 weeks follow up period)
Change of dystrophin expression rate in muscle tissues from the baseline assessment | At 37 weeks (1 week after from 36 weeks treatment period)

SECONDARY OUTCOMES:
North Star Ambulatory Assessment | At 36 weeks
Timed test (6MWT, time to walk/run 10 meters, time to climb/descent four steps, time to rise from the floor) | At 36 weeks
Muscle strength (MMT, QMT) | At 36 weeks
Dairy activities | At 36 weeks
Biomarkers (CK, ALD) | At 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Takeshima, MD, PhD, Principal Investigator — Hyogo Medical University; Hirofumi Komaki, MD, PhD, Study Director — National center of neurology and psychiatry, department of child neurology, Muscular disease center
Locations (4):
- Japan (4):
  - Kobe university hospital, department of pediatrics, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - National center of neurology and psychiatry, Kodaira, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku, Tokyo